CLINICAL TRIAL: NCT00754338
Title: Evaluation of Disinfecting Solutions and Protein Remover With a Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Desmond Fonn, MOptom., Centre for Contact Lens Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: P/279/07/L
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Ametropia
Keywords: comfort; wetability; protein deposit; lipid deposit
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase1 - Arm 1 (Active Comparator)
  Interventions: Drug: Alcon Opti-Free® RepleniSH® with Supraclens®; Drug: Alcon Opti-Free® RepleniSH®
- Phase1 - Arm 2 (Active Comparator)
  Interventions: Drug: Alcon Opti-Free® RepleniSH® with Supraclens®; Drug: Alcon Opti-Free® RepleniSH®
- Phase 2 - Arm 1 (Active Comparator)
  Interventions: Drug: Alcon Opti-Free® RepleniSH® with Supraclens®; Drug: B&L ReNu MultiPlus™
- Phase 2 - Arm 2 (Active Comparator)
  Interventions: Drug: Alcon Opti-Free® RepleniSH® with Supraclens®; Drug: B&L ReNu MultiPlus™

INTERVENTIONS:
Drug: Alcon Opti-Free® RepleniSH® with Supraclens® — Marketed Multipurpose Disinfecting Care System + Marketed contact lens protein remover
Drug: Alcon Opti-Free® RepleniSH® — Marketed Multipurpose Disinfecting Care System
  Arms: Phase1 - Arm 1; Phase1 - Arm 2
Drug: B&L ReNu MultiPlus™ — Marketed Multipurpose Disinfecting Care Systems
  Arms: Phase 2 - Arm 1; Phase 2 - Arm 2

SUMMARY:
The purpose of this study is to determine if reduced lens deposits and increased comfort can be achieved by using Multipurpose disinfecting solutions (MPDS) in a no-rub format but in conjunction with an intensive cleaner, rather than using MPDS in a rub format.

DETAILED DESCRIPTION:
The purpose of this study is to determine if reduced lens deposits and increased comfort can be achieved by using Multipurpose disinfecting solutions (MPDS) in a no-rub format but in conjunction with an intensive cleaner, rather than using MPDS in a rub format by observing changes within the cornea and collecting subjective ratings.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer.
* Has read, understood and signed an information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is correctable to a visual acuity of 6/9 or better (in each eye) with their habitual vision correction.
* Has clear corneas and no active ocular disease.
* Has had an ocular examination in the last two years.
* Is a current soft lens wearer, replacing their lenses every two weeks to one month.
* Has a distance contact lens prescription between +6.00D to -10.00 DS and can be successfully fit with the study lens.
* Has astigmatism less than or equal to -1.00 DC.

Exclusion Criteria:

* Has any signs or symptoms of dry eye.
* Has any clinically significant blepharitis.
* Has undergone corneal refractive surgery.
* Is aphakic.
* Has any active ocular disease.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that may affect ocular health.
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
* Is pregnant or lactating.
* Is participating in any other type of clinical or research study.
* Currently wears daily disposable lenses.
* Currently wears lenses on an extended wear basis.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, MOptom, Study Chair — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, School of Optometry, University of Waterloo., Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started January 2008 at CCLR (Study completed July 2008)
Pre-assignment Details: Phase 1 - 38 participants enrolled, Phase 2 - 38 participants enrolled. For both Phase 1 and 2 a washout period of at least one day, during which time participants wore spectacles and no contact lenses.
Groups:
- Ph1: 1st-RepleniSH(No-rub) & Supraclens, 2nd RepleniSH(Rub): Phase 1 - Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) with 'no lens rub' and Supraclens® (Daily protein remover) first, and Alcon RepleniSH™ 'with lens rub' second. Participants wore PureVision lenses on a daily wear basis for at least eight to ten hours per day and at least six days per week for the duration of the study.
- Ph1: 1st-RepleniSH(Rub), 2nd-RepleniSH(No-rub) & Supraclens: Phase 1 - Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) 'with lens rub' first, and Alcon RepleniSH™ with 'no lens rub' and Supraclens® (Daily protein remover) second. Participants wore PureVision lenses on a daily wear basis for at least eight to ten hours per day and at least six days per week for the duration of the study.
- Ph2: 1st-RepleniSH(No-rub)&Supraclens, 2nd ReNUMultiplus(Rub): Phase 2 - Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) with 'no lens rub' and Supraclens® (Daily protein remover) first, and B&L ReNu MultiPlus™ (Contact lens cleaning and disinfecting solution) 'with lens rub' second. Participants wore PureVision lenses on a daily wear basis for at least eight to ten hours per day and at least six days per week for the duration of the study.
- Ph2: 1st-ReNu Multiplus(Rub), 2nd RepleniSH(No-rub)&Supraclens: Phase 2 - B&L ReNu MultiPlus™ (Contact lens cleaning and disinfecting solution) 'with lens rub' first, and Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) with 'no lens rub' and Supraclens® (Daily protein remover) second. Participants wore PureVision lenses on a daily wear basis for at least eight to ten hours per day and at least six days per week for the duration of the study.
Period: First Intervention for Phase1&Phase2
Arm/Group | Ph1: 1st-RepleniSH(No-rub) & Supraclens, 2nd RepleniSH(Rub) | Ph1: 1st-RepleniSH(Rub), 2nd-RepleniSH(No-rub) & Supraclens | Ph2: 1st-RepleniSH(No-rub)&Supraclens, 2nd ReNUMultiplus(Rub) | Ph2: 1st-ReNu Multiplus(Rub), 2nd RepleniSH(No-rub)&Supraclens
Started | 17 | 21 | 19 | 19
Completed | 17 | 18 | 16 | 19
Not Completed | 0 | 3 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 0
Period: Second Intervention for Phase1&Phase2
Arm/Group | Ph1: 1st-RepleniSH(No-rub) & Supraclens, 2nd RepleniSH(Rub) | Ph1: 1st-RepleniSH(Rub), 2nd-RepleniSH(No-rub) & Supraclens | Ph2: 1st-RepleniSH(No-rub)&Supraclens, 2nd ReNUMultiplus(Rub) | Ph2: 1st-ReNu Multiplus(Rub), 2nd RepleniSH(No-rub)&Supraclens
Started | 17 | 18 | 16 | 19
Completed | 17 | 17 | 16 | 18
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ph1: RepleniSH(No-rub) & Supraclens: Phase 1 - Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) with 'no lens rub' and Supraclens® (Daily protein remover) group.
- Ph1: RepleniSH(Rub): Phase 1 - Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) 'with lens rub' group.
- Ph2: RepleniSH(No-rub) & Supraclens: Phase 2 - Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) with 'no lens rub' and Supraclens® (Daily protein remover) group.
- Ph2: ReNu Multiplus(Rub): Phase 2 - B&L ReNu MultiPlus™ (Contact lens cleaning and disinfecting solution) 'with lens rub' group.
- Total: Total of all reporting groups
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub) | Total
Number analyzed (Participants) | 17 | 21 | 19 | 19 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 19 | 19 | 76
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (11) | 21 (3) | 30 (9) | 24 (7) | 26 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 17 | 14 | 61
  Male | 4 | 4 | 2 | 5 | 15
Region of Enrollment [Number; unit: participants]
  Canada | 17 | 21 | 19 | 19 | 76

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Subjective comfort ratings on analog scale (0= very poor comfort; 100= excellent comfort), self report by subject based on single criterion 'comfort'.
Time Frame: 4 weeks
Population: analysis was per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Ph1: RepleniSH(No-rub) & Supraclens: Phase 1 - Comfort data for Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) with 'no lens rub' and Supraclens® (Daily protein remover) group.
- Ph1: RepleniSH(Rub): Phase 1 - Comfort data for Alcon RepleniSH™ (Contact lens cleaning and disinfecting solution) 'with lens rub' group
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Units on a scale | 86 (13) | 86 (15) | 87 (14) | 86 (14)

2. Secondary Outcome: Dryness
Description: Subjective dryness ratings on analog scale (0= very dry; 100= not dry at all), self report by subject based on single criterion 'dryness'.
Time Frame: 4 weeks
Population: analysis was per protocol
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Units on a Scale | 85 (14) | 86 (16) | 85 (15) | 85 (15)

3. Secondary Outcome: Subjective Vision
Description: Subjective vision ratings on analog scale (0= poor vision; 100= excellent vision), self report by subject based on single criterion 'vision'.
Time Frame: 4 weeks
Population: analysis was per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Units on a scale | 89 (12) | 89 (13) | 90 (11) | 90 (11)

4. Secondary Outcome: Corneal Staining
Description: Grading based on Type (0=None; 100=patch)and extent of staining (0=None; 100= Entire corneal region). Final value is Type multiplied by Extent.
  Corneal staining is a test that uses an orange dye (fluorescein) and a blue light to detect damage to the cornea (front surface of eye) from minor abrasions.
  A strip of blotting paper containing the dye was touched to the eyelid margin. Upon blinking, the dye spreads and coats the front surface of the eye along with the tear film covering the surface of the cornea. The investigator then rated the size, location and shape of the staining.
Time Frame: 4 weeks
Population: analysis was per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Units on a scale | 47 (111) | 55 (113) | 52 (108) | 322 (479)

5. Primary Outcome: Lens Wettability
Description: Subjective grading of contact lens surface wettability by investigator (0=excellent; 4=severely reduced).
Time Frame: 4 weeks
Population: analysis was per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Units on a scale | 0.71 (0.49) | 0.72 (0.38) | 0.92 (0.68) | 1.21 (0.69)

6. Primary Outcome: Lens Deposits
Description: Subjective grading of contact lens surface deposits by investigator (0=no deposits; 4=severe deposits).
Time Frame: 4 weeks
Population: analysis was per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub)
Number analyzed (Participants) | 34 | 34 | 34 | 34
Units on a scale | 0.51 (0.34) | 0.54 (0.47) | 0.62 (0.43) | 0.93 (0.66)

ADVERSE EVENTS:
Time Frame: One business day to Office of Research Ethics
Description: No adverse events were reported for this study.
Arm/Group | Ph1: RepleniSH(No-rub) & Supraclens | Ph1: RepleniSH(Rub) | Ph2: RepleniSH(No-rub) & Supraclens | Ph2: ReNu Multiplus(Rub)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days